CLINICAL TRIAL: NCT01505855
Title: Serological Response to Pneumococcal Vaccination in Crohn's Disease: A Prospective Multicenter Study
Brief Title: Efficacy Study of Pneumococcal Vaccination in Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Wonju Severance Christian Hospital (Other); Seoul National University Hospital (Other); Asan Medical Center (Other); Soonchunhyang University Hospital (Other); Ewha Womans University (Other); Kosin University Gospel Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Inje University (Other); The Catholic University of Korea (Other); Keimyung University Dongsan Medical Center (Other); Korea University (Other); Wonkwang University (Other); Severance Hospital (Other); Konkuk University Hospital (Other)
Responsible Party: Principal Investigator, Chang Kyun Lee, Assistant Professor, Kyunghee University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CD vaccination 1.2
Record Dates: First submitted 2012-01-02; First posted 2012-01-09 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Pneumococcal vaccination
MeSH Terms: conditions — Crohn Disease | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- anti-TNF only (Experimental): Crohn's disease, on an anti-TNF agent [infliximab or adalimumab] only
  Interventions: Drug: 23-valent polysaccharide pneumococcal vaccine
- Combined immunosuppression (Experimental): Crohn's disease, on combined immunosuppression (both anti-TNF agent and immunomodulator [azathioprine or 6-MP])
  Interventions: Drug: 23-valent polysaccharide pneumococcal vaccine
- Immunomodulator only (Experimental): Crohn's disease, on an immunomodulator only
  Interventions: Drug: 23-valent polysaccharide pneumococcal vaccine
- Non-immunosuppression (Experimental): Crohn's disease, not on immunosuppressive medications (5-ASA only: control arm)
  Interventions: Drug: 23-valent polysaccharide pneumococcal vaccine

INTERVENTIONS:
Drug: 23-valent polysaccharide pneumococcal vaccine — 23-valent polysaccharide pneumococcal vaccine (PSV-23 vaccine) 0.5mL single intramuscular injection
  Other Names: Pneumovax

SUMMARY:
A growing number of patients with Crohn's disease are treated with immunosuppressive agents, such as anti-tumor necrosis factor blockers and immunomodulators. Several recent studies have indicated that immunosuppressive treatment may impair the immunological response to pneumococcal vaccination in patients with inflammatory bowel disease (Crohn's disease and Ulcerative colitis). One of weaknesses in the previous studies did not focus on specific disease, such as Crohn's disease. In addition, predictive factors affecting impaired response following pneumococcal vaccination have not clearly evaluated in patients with Crohn's disease. In this study, patients with Crohn's disease will be assessed for serological response to pneumococcal vaccination. Further, potential predictive factors that impact on vaccination outcomes and adverse events related to vaccination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Informed consent
* Patients who had a definitive diagnosis of Crohn's disease for more than 6 months (documented by the standard clinical, radiographic, endoscopic, and histopathologic criteria)

Exclusion Criteria:

* Hypersensitivity to any component of the pneumococcal vaccine
* Known allergy to pneumococcal vaccination
* Patients who treated with glucocorticoids (prednisolone > 20 mg/day equivalent for 2 weeks or more, and within 3 months of stopping
* Patients who inoculate another vaccine in the past 4 weeks
* Significant protein calorie malnutrition
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, infectious, neurologic or cerebral disease
* Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he/she were to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Serological response rates | 4 weeks
  Serological response rates, defined by number of patients showing adequate response to pneumococcal vaccination (at least a 2-fold increase in antipneumococcal antibodies in the serum compared with baseline)

SECONDARY OUTCOMES:
Safety assessment of the vaccine | 8 weeks
  adverse events related to vaccine administration, including worsening of Crohn's disease activity by changes in Harvey-Bradshaw index (HBI) and inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Soo Kim, MD, PhD, Study Chair — Yonsei University
Locations (15):
- South Korea (15):
  - Yonsei University: Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Kosin University Gospel Hospital, Busan
  - Soonchunhyang University, Cheonan
  - Keimyung University; Dongsan Hospital, Daegu
  - Wonkwang University, Iksan
  - Kyung Hee University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University, Seoul
  - Ewha Womans University, Seoul
  - Inje University; Seoul Paik Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Korea University; Ansan Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University; Severance Hospital, Seoul
  - The Catholic University of Korea; St. Vincent's Hospital, Suwon

REFERENCES:
- [Background] Melmed GY, Agarwal N, Frenck RW, Ippoliti AF, Ibanez P, Papadakis KA, Simpson P, Barolet-Garcia C, Ward J, Targan SR, Vasiliauskas EA. Immunosuppression impairs response to pneumococcal polysaccharide vaccination in patients with inflammatory bowel disease. Am J Gastroenterol. 2010 Jan;105(1):148-54. doi: 10.1038/ajg.2009.523. Epub 2009 Sep 15. PMID 19755964
- [Background] Fiorino G, Peyrin-Biroulet L, Naccarato P, Szabo H, Sociale OR, Vetrano S, Fries W, Montanelli A, Repici A, Malesci A, Danese S. Effects of immunosuppression on immune response to pneumococcal vaccine in inflammatory bowel disease: a prospective study. Inflamm Bowel Dis. 2012 Jun;18(6):1042-7. doi: 10.1002/ibd.21800. Epub 2011 Jun 14. PMID 21674732
- [Background] Wasan SK, Coukos JA, Farraye FA. Vaccinating the inflammatory bowel disease patient: deficiencies in gastroenterologists knowledge. Inflamm Bowel Dis. 2011 Dec;17(12):2536-40. doi: 10.1002/ibd.21667. Epub 2011 Apr 28. PMID 21538710